CLINICAL TRIAL: NCT01852357
Title: A Placebo-Control Evaluation of Neurofeedback Efficacy in Adults With ADHD
Brief Title: An Evaluation of Neurofeedback Efficacy in Adults With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Wilmington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: R15AT007226 (NIH)
Record Dates: First submitted 2013-04-26; First posted 2013-05-13 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2014-06

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham control (Sham Comparator): This group will receive 12 sham neurofeedback sessions in which the feedback is based on pre-recorded data.
  Interventions: Other: Sham Neurofeedback
- Neurofeedback (Experimental): The intervention will be 24 sessions of beta/SMR neurofeedback.
  Interventions: Other: Neurofeedback

INTERVENTIONS:
Other: Neurofeedback — The intervention will be 24 sessions of beta/sensorimotor rhythm (SMR) neurofeedback.
  Other Names: EEG biofeedback
  Arms: Neurofeedback
Other: Sham Neurofeedback — Feedback generated by data not associated with the current participant.
  Arms: Sham control

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of neurofeedback training (NFB) on objective measurements of attention in young adults with ADHD. The secondary objectives are to evaluate neurofeedback effects on self-report measures of attention, ADHD symptoms, and to identify electroencephalogram (EEG) markers of ADHD and neurofeedback efficacy. The study is a double-blind, placebo controlled clinical trial to test the efficacy and safety of EEG neurofeedback in individuals 18-40 years of age with attention deficit hyperactivity disorder (ADHD). Attention will be evaluated at baseline, after 12 and 24 training sessions (an average of 4 and 8 weeks, respectively), and 4 weeks after the last neurofeedback session. The primary outcome will be change from baseline on the Attention Performance Index (API) variable of the Test of Variables of Attention (TOVA) a standardized, well-normed, computerized test of attention, after 12 neurofeedback or sham training sessions (and average of 4 weeks). Secondary outcomes will be change from baseline on other TOVA variables after 12 and 24 sessions (an average of 4 and 8 weeks, respectively), at 4 weeks post-training follow-up, and changes from baseline at each time point on the Adult Self Report Scale (ASRS) and Mindful Awareness and Attention Scale (MAAS). EEG data collected during TOVA attention testing at baseline will be used to model EEG differences between ADHD and non-ADHD participants. Additional EEG data collected during the TOVA at midpoint (average of 4 weeks), after 24 NFB sessions (average of 8 weeks), and 4 weeks post-NFB will be used to develop statistical models to use as indicators of neurofeedback efficacy

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 40 years old.
* ADHD participants must have a previous diagnosis of ADHD (inattentive or mixed type) by a licensed psychologist or psychiatrist.
* ADHD participants must have scores on the Adult Self-Report Scale V1.1 (ASRS; (Kessler et al. 2005)) > 24.
* ADHD participants must have TOVA API z score < 0.
* Ability to understand study procedures and to comply with them for the entire length of the study.
* Men and women of reproductive capability will be enrolled. Contraception is not necessary or required.

Exclusion Criteria:

* A history of psychiatric disorder.
* Scores in clinical ranges on the Beck Depression Inventory II (20 or above) or Beck Anxiety Inventory (16 or above).
* A history of seizures.
* Known neurological disorders.
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of individual to give written informed consent.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Attention Performance Index of the Test of Variables of Attention | After 12 neurofeedback or sham sessions (an average of 4 weeks).
  The primary outcome will be change from baseline on the Attention Performance Index (API) variable of the Test of Variables of Attention (TOVA) a standardized, well-normed, computerized test of attention, after 12 neurofeedback or sham training sessions (an average of 4 weeks).

SECONDARY OUTCOMES:
Test of Variables of Attention | after 12 (average 4 weeks) and 24 sessions (average 8 weeks) and 1 month followup
  Secondary outcomes will be change from baseline on other TOVA variables after 12 and 24 sessions (4 and 8 weeks on average, respectively), at 4 weeks post-training follow-up

OTHER OUTCOMES:
Adult Self-Report Scale | after 12 and 24 sessions (average of 4 and 8 weeks, respectively), 1 month followup
  A self report survey of ADHD symptoms.
Mindful Awareness and Attention Scale | after 12 and 24 sessions (average of 4 and 8 weeks, respectively) and 1 month followup
  A self report scale that assesses mindful attention and awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Julian R Keith, Ph.D, Principal Investigator — University of North Carolina, Wilmington
Locations (1):
- Department of Psychology, UNC Wilmington, Wilmington, North Carolina, United States